CLINICAL TRIAL: NCT07324512
Title: Determination of the Minimum Effective Volume of Crystalloid Co-Loading for Preventing Spinal Anesthesia-Induced Hypotension in Cesarean Section: A Biased Coin Design Study
Brief Title: Minimum Effective Volume of Crystalloid Co-Loading to Prevent Spinal Anesthesia-Induced Hypotension in Cesarean Section
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2508-038-1665
Record Dates: First submitted 2025-12-14; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-10

CONDITIONS: Spinal Induced Hypotension in Cesarean Delivery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Crystalloid Co-Loading (Experimental): Participants undergo spinal anesthesia for elective cesarean delivery. Immediately after intrathecal injection, a predefined volume of balanced crystalloid (co-loading) is infused over ~10 minutes while a prophylactic phenylephrine infusion is initiated per protocol. The crystalloid volume for each successive participant is adjusted using a biased-coin up-and-down algorithm to identify the minimum effective volume that prevents spinal-anesthesia-induced hypotension in ≥90% of patients (MEV90, mL/kg). Blood pressure is monitored frequently; rescue phenylephrine and/or fluids are permitted to maintain predefined blood pressure ranges. Maternal adverse events and neonatal outcomes are recorded through postoperative day 2.
  Interventions: Other: Intravenous Crystalloid Co-Loading

INTERVENTIONS:
Other: Intravenous Crystalloid Co-Loading — Balanced crystalloid is infused intravenously immediately after intrathecal injection as a co-load. A predefined volume (mL/kg) is administered over ~10 minutes. The volume for successive participants is adapted by a biased-coin up-and-down algorithm to estimate the minimum effective volume (MEV90) that prevents spinal-anesthesia-induced hypotension. Rescue fluids are allowed per protocol.

SUMMARY:
The goal of this clinical trial is to find the minimum effective volume of IV crystalloid that should be given with phenylephrine to prevent hypotension caused by spinal anesthesia in healthy, term pregnant adults having elective cesarean delivery.

The main questions are:

What is the minimum effective volume (MEV90, mL/kg) of crystalloid co-loading that prevents spinal-anesthesia-induced hypotension in ≥90% of participants?

What maternal side effects and newborn outcomes occur with this strategy (e.g., nausea/vomiting, need for extra vasopressors, total fluids/blood loss, Apgar scores, and umbilical cord blood gases)?

There is no separate comparison group; this is a single-arm, adaptive dose-finding study.

Participants will:

Receive a predefined volume of IV crystalloid over ~10 minutes during spinal anesthesia while phenylephrine is infused. Have blood pressure and symptoms monitored; receive rescue treatment if needed. Allow the next participant's fluid volume to be adjusted based on whether hypotension occurred (biased-coin design). Be followed through postoperative day 2 for maternal and newborn outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant adults ≥19 years scheduled for elective cesarean delivery under spinal anesthesia
* Term pregnancy (≥37 weeks' gestation)

Exclusion Criteria:

* Emergency cesarean delivery
* Hypertensive disorders of pregnancy (preeclampsia/eclampsia) or hypertension
* Multiple gestation
* Body weight <50 kg or BMI >35 kg/m²
* Renal impairment or eGFR ≤90 mL/min/1.73 m²
* Heart failure or other heart disease
* History of bronchial asthma or other pulmonary disease

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-27 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Minimum Effective Volume (MEV90) of Intravenous Crystalloid Co-Loading (mL/kg) | From intrathecal injection (start of spinal anesthesia) to end of surgery
  The smallest crystalloid co-loading dose (mL/kg) that prevents spinal-anesthesia-induced hypotension in ≥90% of participants when given with prophylactic phenylephrine.

SECONDARY OUTCOMES:
Incidence of intraoperative hypotension (mmHg) | From intrathecal injection to end of surgery
  Hypotension is defined as a drop in systolic blood pressure (SBP) to < 80% of the participant's baseline SBP (mmHg). Baseline SBP is the mean of the last three ward SBP measurements obtained before operating room admission.
Incidence of intraoperative hypertension (mmHg) | From intrathecal injection to end of surgery
  Hypertension is defined as any occurrence of systolic blood pressure (SBP) > 120% of baseline SBP (mmHg) after spinal anesthesia. Baseline SBP is the mean of the last three ward SBP measurements obtained before operating room admission.
Additional bolus phenylephrine requirement | From intrathecal injection to end of surgery
  Administration of rescue phenylephrine bolus in addition to the protocolized prophylactic phenylephrine infusion to treat or prevent hypotension after spinal anesthesia. Hypotension is defined as SBP < 80% of baseline SBP (mmHg) or MAP < 65 mmHg. Baseline SBP is the mean of the last three ward SBP measurements obtained before operating room admission. When hypotension occurs, phenylephrine 100 µg is administered as an IV bolus to restore blood pressure. The outcome is recorded as number of phenylephrine boluses.
Total Phenylephrine Dose (µg) | From intrathecal injection to end of surgery
  Total intraoperative phenylephrine dose administered after spinal anesthesia, defined as the sum of the prophylactic infusion dose and all rescue bolus doses. he prophylactic infusion starts at 1,500 µg/h and the infusion rate is reduced if systolic blood pressure (SBP) exceeds 120% of baseline SBP (mmHg). Baseline SBP is the mean of the last three ward SBP measurements obtained before operating room admission. Rescue bolus protocol: phenylephrine 100 µg IV per hypotensive episode (SBP < 80% of baseline SBP [mmHg] or MAP < 65 mmHg), repeated as needed. Dose will be abstracted from the anesthesia record (infusion rate × time plus boluses) and summarized in micrograms (µg).
Estimated blood loss (mL) | From skin incision to end of surgery
  Calculated as (suction canister volume - irrigation volume) + gravimetric estimate of soaked sponges/drapes (1 g ≈ 1 mL). For cesarean delivery, amniotic fluid is excluded.
Incidence of Maternal Nausea Associated With Hypotension | From intrathecal injection to end of surgery
  Occurrence of nausea temporally associated with hypotension after spinal anesthesia. Recorded as yes/no (≥1 episode) and number of episodes.
Incidence of Maternal Vomiting Associated With Hypotension | From intrathecal injection to end of surgery
  Occurrence of vomiting temporally associated with hypotension after spinal anesthesia. Recorded as yes/no (≥1 episode) and number of emetic events.
Incidence of Maternal Dizziness/Lightheadedness Associated With Hypotension | From intrathecal injection to end of surgery
  Occurrence of dizziness/lightheadedness temporally associated with hypotension after spinal anesthesia. Recorded as yes/no (≥1 episode) and number of episodes.
Neonatal Apgar score at 1Minute | At 1 minute after birth
  The Apgar score (range 0-10) assessed 1 minute after birth by clinical staff according to standard practice. It is the sum (0-2 each) of heart rate, respiratory effort, muscle tone, reflex irritability, and skin color. Recorded as the total score (0-10) and, if available, the five component scores.
Neonatal Apgar Score at 5 Minutes | At 5 minutes after birth
  The Apgar score (range 0-10) assessed 5 minutes after birth by clinical staff according to standard practice. It is the sum (0-2 each) of heart rate, respiratory effort, muscle tone, reflex irritability, and skin color. Recorded as the total score (0-10) and, if available, the five component scores.
Umbilical Arterial pH | At delivery (immediately after birth)
  Umbilical cord arterial blood gas pH obtained immediately after birth from a double-clamped cord segment and analyzed per routine laboratory practice.
Umbilical Arterial Base Excess (mmol/L) | At delivery (immediately after birth)
  Umbilical cord arterial blood gas base excess measured immediately after birth from a double-clamped cord segment, processed per routine laboratory practice.
Pulmonary edema | Through postoperative day 2
  New-onset pulmonary edema within 48 hours after surgery, defined by physician diagnosis supported by clinical findings (e.g., dyspnea, crackles) and/or objective evidence (e.g., new supplemental oxygen requirement or SpO₂ ≤ 92% on room air, chest imaging consistent with interstitial/alveolar edema). Record as yes/no (≥1 event).
Clinically Significant Generalized Edema | Through postoperative day 2
  Generalized pitting edema present within 48 hours after surgery, defined by ≥1 of the following objective criteria (excluding localized, surgical-site-limited edema):
  (A) Physical exam: pitting grade ≥2+ in ≥2 anatomic regions (e.g., bilateral pretibial/ankle, hands/forearms, sacral, or periorbital), using the standard indentation scale - 2+: ~4 mm pit, brief rebound; 3+: ~6 mm pit, 10-60 s rebound; 4+: ~8 mm pit, >60 s rebound.
  (B) Anthropometry: body weight increase ≥2% (or ≥2 kg) from the preoperative baseline or bilateral mid-calf circumference increase ≥2 cm from baseline.
  (C) Therapeutic criterion: initiation or escalation of diuretic therapy (e.g., IV/PO loop diuretic) for generalized edema as judged by the treating clinician.
  Recorded as yes/no (≥1 criterion met)
Acute Heart Failure | Through postoperative day 2
  New diagnosis of acute heart failure within 48 hours after surgery, characterized by symptoms/signs (e.g., dyspnea, orthopnea, pulmonary congestion), objective evidence (e.g., chest radiographic congestion, elevated BNP/NT-proBNP if available, or echocardiographic findings), and requirement for treatment (e.g., IV diuretics, vasodilators, inotropes, or noninvasive ventilation). Record as yes/no (≥1 event).